CLINICAL TRIAL: NCT01675232
Title: A Randomized, Investigator-Blinded Study Comparing the Efficacy of Two Topical Steroid Application Regimens in Pediatric Patients With Atopic Dermatitis
Brief Title: A Study Comparing the Efficacy of Two Topical Steroid Application Regimens in Pediatric Patients With Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Richard Antaya, Professor of Dermatology and Pediatrics, Yale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIC-1206010366
Record Dates: First submitted 2012-08-02; First posted 2012-08-29 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; Topical corticosteroid; Pediatric; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Soak and smear (Active Comparator): Application of hydrocortisone 2.5% ointment or triamcinolone acetonide 0.1% ointment immediately to wet skin once a day and dry skin once a day.
  Interventions: Other: Soak and smear
- Dry smear (Active Comparator): Application of hydrocortisone 2.5% ointment or triamcinolone acetonide 0.1% ointment to dry skin twice a day.
  Interventions: Other: Dry Smear

INTERVENTIONS:
Other: Soak and smear — Corticosteroid ointment applied to wet skin once a day and dry skin once a day.
  Arms: Soak and smear
Other: Dry Smear — Corticosteroid ointment applied to dry skin twice a day.
  Arms: Dry smear

SUMMARY:
The purpose of this study is to investigate the efficacy of two different corticosteroid ointment application regimens for the treatment of eczema (atopic dermatitis).

ELIGIBILITY:
Inclusion Criteria:

* Meet the clinical criteria for the diagnosis of atopic dermatitis
* Have disease over at least 5% of their total body surface area.
* Less than 18 years of age.
* Families able to comprehend written instructions in English and able to complete questionnaires with assistance if needed.
* Parents/guardians able to understand and willing to sign a parental permission form.
* Children between the ages of 7-17 years willing to sign an age-appropriate assent form.

Exclusion Criteria:

* Patients who are allergic or intolerant of the topical medications employed in this study.
* Lack of follow-up after initial visit or regimen noncompliance.
* Patients who do not have access to a bathtub.

Ages: 2 Weeks to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Efficacy of corticosteroid application regimen as assessed by the Eczema Area and Severity Index (EASI) | 2 weeks

SECONDARY OUTCOMES:
Effect of corticosteroid ointment application regimens on serum cortisol | 2 weeks after application of topical corticosteroids
Frequency of atopic dermatitis flares in the 3 months following the two-week treatment regimen | 3 months
Adverse effects associated with each corticosteroid application regimen | 3 months
  Characterize and quantify adverse effects associated with each corticosteroid application regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Antaya, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States